CLINICAL TRIAL: NCT03471572
Title: A Non-interventional, Multicentre Study to Assess Prevalence of BRCA1 and BRCA2 Mutation Among Ovarian, Primary Peritoneal and Fallopian Tube Cancer Patients in India
Brief Title: Study to Assess Prevalence of BRCA1 and BRCA2 Mutation Among Ovarian, Primary Peritoneal and Fallopian Tube Cancer Patients in India
Acronym: BRCA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0818R00001
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Ovarian Cancer
Keywords: BRCA, ovarian cancer, fallopian tube cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Ovarian Cancer

SUMMARY:
This is a non-interventional, cross-sectional, multicentre, observational study planned to be conducted at 15 sites across all geographical regions of India. The study targets to enrol 240 patients with approximately 16 patients from each site. Written approval of Independent Ethics Committee (IEC)/ Institutional Review Board (IRB) and written informed consent from willing patients will be obtained prior to the start of the study.

DETAILED DESCRIPTION:
This is a non-interventional, cross-sectional, multicentre, observational study to be conducted at 15 sites from different geographical regions across India. The study targets to enrol 240 patients with nearly 16 patients per site over 6 months. The study will enrol females with diagnosis of ovarian, primary peritoneal, or fallopian tube cancer. No study medication will be prescribed or administered as a part of study procedure.

The study will start only after obtaining written approval of Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and written informed consent of the patient.

The study will start only after obtaining written approval of Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and written informed consent of the patient. Eligible patients will undergo physical examination and data of demographics, vital signs, present/ past history of illness, family history of breast/ovarian cancer, current and previous chemotherapy regimen and current medication will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provide written informed consent
2. Female ≥ 18 years of age
3. Previously or newly diagnosed ovarian, primary peritoneal, or fallopian tube cancer patients.

Exclusion Criteria:

1. Patient with any medical condition that, in the opinion of the investigator, would interfere with safe completion of the study

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously or newly diagnosed ovarian, primary peritoneal, or fallopian tube cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
BRCA1 or BRCA2 mutation positive status | 1 day
  ENIGMA (Evidence-based Network for the Interpretation of Germline Mutant Alleles)

SECONDARY OUTCOMES:
Association between histopathological type and BRCA 1/BRCA 2 mutation positive status | 1 Day
  Frequency of different histopathological type and BRCA 1/BRCA 2 mutation positive status will be presented.

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Research Site, Bangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Delhi, New Delhi
  - Research Site, Hyderabad, Telangana
  - Research Site, Kolkata, West Bengal

REFERENCES:
- See also: Redacted_csr_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0818R00001&attachmentIdentifier=1d220cab-775e-4bad-bee4-a1d76d7f4c1f&fileName=redacted_csr_synopsys_BRCA_study.pdf&versionIdentifier=